CLINICAL TRIAL: NCT03750565
Title: A Multiple Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TD-1473 in Healthy Adult Japanese Subjects
Brief Title: Multiple Dose Ethnobridging PK Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0176
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Inflammatory Bowel Diseases; IBD
Keywords: Healthy Japanese Subjects; Healthy Caucasian Subjects; Ethnobridging
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Japanese subjects will receive oral doses of either TD-1473 - Dose A or placebo (15 healthy Japanese subjects randomized 3:1 to 12 active and 3 placebo) once daily (QD) for 14 consecutive days.
  Interventions: Drug: TD-1473 - Dose A; Drug: Placebo
- Cohort 2 (Experimental): Japanese subjects will receive oral doses of either TD-1473 - Dose B or placebo (15 healthy Japanese subjects randomized 3:1 to 12 active and 3 placebo) once daily (QD) for 14 consecutive days.
  Interventions: Drug: TD-1473 - Dose B; Drug: Placebo
- Cohort 3 (Experimental): Caucasian subjects will receive oral doses of either TD-1473 - Dose B or placebo (15 healthy Caucasian subjects randomized 3:1 to 12 active and 3 placebo) once daily (QD) for 14 consecutive days.
  Interventions: Drug: TD-1473 - Dose B; Drug: Placebo
- Cohort 4 (Experimental): Japanese subjects will receive oral doses of either TD-1473 - Dose C or placebo (15 healthy Japanese subjects randomized 3:1 to 12 active and 3 placebo) once daily (QD) for 14 consecutive days.
  Interventions: Drug: TD-1473 - Dose C; Drug: Placebo

INTERVENTIONS:
Drug: TD-1473 - Dose A — oral capsule/tablet, QD
  Arms: Cohort 1
Drug: TD-1473 - Dose B — oral capsule/tablet, QD
  Arms: Cohort 2; Cohort 3
Drug: TD-1473 - Dose C — oral capsule/tablet, QD
  Arms: Cohort 4
Drug: Placebo — oral capsule/tablet, QD

SUMMARY:
A Phase 1, double blind, placebo controlled, 4 cohort, multiple dose study in healthy adult Japanese and Caucasian subjects.

ELIGIBILITY:
Inclusion Criteria:

For All subjects:

* Male or female between 18 to 55 years old
* Female subjects must have documentation of a negative serum pregnancy test,
* Female subjects must be either of non-childbearing potential or if of childbearing potential use a highly efficient birth control method
* Male subjects must be vasectomized with documented medical assessment of the surgical success, or use acceptable contraception
* All male subjects must agree to refrain from sperm donation during the study and for at least 7 days after the last dose of study drug.
* Body Mass Index (BMI) 18 to 32 kg/m2, inclusive, and weighs at least 50 kg and less than 90 kg
* Willing and able to give informed consent
* Additional inclusion criteria apply

For Japanese subjects only:

* Subject must have been born in Japan, with 2 Japanese biological parents and 4 Japanese grandparents as confirmed by interview.
* Subject has lived no longer than 10 years outside of Japan.
* Subject had no significant change in lifestyle, including diet, since leaving Japan.

For Caucasian subjects only:

* Subject has 2 Caucasian biological parents and 4 Caucasian grandparents as confirmed by interview.
* Subject has lived no longer than 10 years outside of Europe and/or North America.

Exclusion Criteria:

For all subjects:

* Subject is a female who is pregnant, lactating, breastfeeding, or planning to become pregnant during the study or within 7 days after the last dose of study drug.
* Subject is a male who is planning to father a child during the study or within 7 days after the last dose of study drug.
* Is positive for hepatitis A, B or C, and/or HIV
* Has clinically significant abnormalities in baseline laboratory evaluations
* Subject has a clinically significant abnormal electrocardiogram (ECG)
* Participated in another clinical trial of an investigational drug (or medical device) within 30 days prior to screening or is currently participating in another trial of an investigational drug (or medical device) Additional exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-02-13 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve (AUC0 t) | Day 1 & Day 14
Area under the concentration-time curve (AUC0 24) | Day 1 & Day 14
Area under the concentration-time curve (AUCtau) | Day 1 & Day 14
Maximum observed concentration (Cmax) | Day 1 & Day 14
Maximum observed concentration at steady state (Cmax_ss) | Day 1 & Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- Theravance Biopharma Investigational Site, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No
Theravance Biopharma, Inc. will not be sharing individual de-identified participant data or other relevant study documents.